CLINICAL TRIAL: NCT02586025
Title: A Randomized, Multicenter, Double-Blind, Placebo-Controlled, Phase III Study to Evaluate Pertuzumab in Combination With Docetaxel and Trastuzumab as Neoadjuvant Therapy, and Pertuzumab in Combination With Trastuzumab as Adjuvant Therapy After Surgery and Chemotherapy in Patients With Early-Stage or Locally Advanced HER2-Positive Breast Cancer
Brief Title: Study in Participants With Early-Stage or Locally Advanced Human Epidermal Growth Factor Receptor (HER) 2-Positive Breast Cancer to Evaluate Treatment With Trastuzumab Plus (+) Pertuzumab + Docetaxel Compared With Trastuzumab + Placebo + Docetaxel
Acronym: PEONY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YO28762
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Surgical Procedures, Operative; Docetaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Trastuzumab, Pertuzumab, and Chemotherapy (Experimental): Prior to surgery: trastuzumab, pertuzumab, and docetaxel for 4 cycles (1 cycle = 21 days). After surgery/chemotherapy with 5-fluorouracil, epirubicin, and cyclophosphamide (FEC): trastuzumab and pertuzumab up to 1 year total.
  Interventions: Drug: FEC Chemotherapy; Procedure: Surgery; Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Trastuzumab, Placebo, and Chemotherapy (Experimental): Prior to surgery: trastuzumab, placebo, and docetaxel for 4 cycles (1 cycle = 21 days). After surgery/FEC chemotherapy: trastuzumab and placebo up to 1 year total.
  Interventions: Drug: FEC Chemotherapy; Procedure: Surgery; Drug: Docetaxel; Drug: Placebo; Drug: Trastuzumab

INTERVENTIONS:
Drug: FEC Chemotherapy — Fluorouracil 500-600 milligrams per square meter (mg/m2), epirubicin 90-120 mg/m2, and cyclophosphamide 500-600 mg/m2 by intravenous (IV) infusion every 3 weeks for three cycles (Cycles 5-7). FEC chemotherapeutic agents will be administered following surgery on Day 1 of each specified cycle.
Procedure: Surgery — All participants who are eligible for surgery will undergo surgery and have their pathologic response evaluated.
Drug: Docetaxel — Docetaxel IV infusion in 3-week cycles. Neoadjuvant treatment: 75 mg/m2 for Cycles 1-4.
Drug: Pertuzumab — Pertuzumab IV infusion in 3-week cycles. Prior to surgery (neoadjuvant treatment): 840 milligrams (mg) loading dose for Cycle 1, followed by 420 mg for Cycles 2-4. After surgery and 3 cycles of FEC chemotherapy (adjuvant treatment): 840 mg loading dose for Cycle 8, followed by 420 mg for Cycles 9-20)
  Other Names: RO4368451
  Arms: Trastuzumab, Pertuzumab, and Chemotherapy
Drug: Placebo — Placebo by IV infusion in 3-week cycles as neoadjuvant treatment (Cycles 1-4)and as adjuvant treatment (Cycles 8-20)
  Arms: Trastuzumab, Placebo, and Chemotherapy
Drug: Trastuzumab — Trastuzumab IV infusion in 3-week cycles. Neoadjuvant treatment: 8 milligrams per kilogram (mg/kg) loading dose for Cycle 1, followed by 6 mg/kg for Cycles 2-4. Adjuvant treatment: 8 mg/kg loading dose for Cycle 8, followed by 6 mg/kg for Cycles 9-20.
  Other Names: RO0452317

SUMMARY:
This is an Asia-Pacific regional, randomized, double-blind, multicenter trial designed to evaluate treatment with trastuzumab + pertuzumab + docetaxel compared with trastuzumab + placebo + docetaxel in chemotherapy-naïve participants with early-stage or locally advanced HER2-positive breast cancer. The anticipated treatment duration is approximately 17 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast carcinoma with a primary tumor size of more than (>) 2 centimeters (cm) by standard local assessment technique
* Breast cancer stage at presentation: early-stage (T2-3, N0-1, M0) or locally advanced (T2-3, N2 or N3, M0; T4, any N, M0)
* HER2-positive breast cancer confirmed by a Sponsor-designated central laboratory and defined as 3+ score by immunohistochemistry in > 10 percent (%) of immunoreactive cells or HER2 gene amplification (ratio of HER2 gene signals to centromere 17 signals equal to or more than [>=] 2.0) by in situ hybridization
* Known hormone receptor status (estrogen receptor and/or progesterone receptor)
* Eastern Cooperative Oncology Group Performance Status equal to or less than (<=) 1
* Baseline left ventricular ejection fracture >= 55% measured by echocardiography (preferred) or multiple gated acquisition scan
* Negative serum pregnancy test

Exclusion Criteria:

* Stage IV metastatic breast cancer
* Inflammatory breast cancer
* Previous anti-cancer therapy or radiotherapy for any malignancy
* History of other malignancy within 5 years prior to screening, except for appropriately-treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Concurrent anti-cancer treatment in another investigational trial, including hormone therapy, bisphosphonate therapy, or immunotherapy
* Major surgical procedure unrelated to breast cancer within 4 weeks prior to randomization or from which the participant has not fully recovered
* Serious cardiac illness or medical condition
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness
* Any abnormalities in liver, kidney or hematologic function laboratory tests immediately prior to randomization
* Sensitivity to any of the study medications, any of the ingredients or excipients of these medications, or benzyl alcohol
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2017-10-23 (Actual); Study Completion 2022-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- China (13):
  - The Affiliated Hospital of Military Medical Sciences(The 307th Hospital of Chinese PLA), Beijing
  - the First Hospital of Jilin University, Changchun
  - Jilin Cancer Hospital, Changchun
  - Fujian Medical University Union Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- South Korea (3):
  - Kyungpook National University Medical Center, Daegu
  - Ajou University Medical Center, Gyeonggi-do
  - Korea University Guro Hospital, Seoul
- Taiwan (4):
  - Taipei Medical University ?Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital; Surgery, Taichung
  - Mackay Memorial Hospital; Dept of Surgery, Taipei
  - Taipei Medical University Hospital, Taipei
- Thailand (3):
  - Bhumibol Adulyadej Hospital; Medicine, Bangkok
  - Srinagarind Hospital, Khon Kaen University; Surgery, Khon Kaen
  - Songklanagarind Hospital; Department of Surgery, Songkhla

REFERENCES:
- [Derived] Shao Z, Pang D, Yang H, Li W, Wang S, Cui S, Liao N, Wang Y, Wang C, Chang YC, Wang H, Kang SY, Seo JH, Shen K, Laohawiriyakamol S, Jiang Z, Li J, Zhou J, Althaus B, Mao Y, Eng-Wong J. Efficacy, Safety, and Tolerability of Pertuzumab, Trastuzumab, and Docetaxel for Patients With Early or Locally Advanced ERBB2-Positive Breast Cancer in Asia: The PEONY Phase 3 Randomized Clinical Trial. JAMA Oncol. 2020 Mar 1;6(3):e193692. doi: 10.1001/jamaoncol.2019.3692. Epub 2020 Mar 12. PMID 31647503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 329 participants with early-stage or locally advanced human epidermal growth factor receptor (HER) 2-positive breast cancer were enrolled in this study at 23 investigative sites in China, Republic of Korea, Taiwan, and Thailand from 14 March 2016 to 14 March 2022.
Groups:
- Pertuzumab, Trastuzumab, and Chemotherapy: Prior to surgery: Participants received trastuzumab, 8 milligrams per kilograms (mg/kg) loading dose in Cycle 1, followed by 6 mg/kg from Cycles 2-4, pertuzumab, 840 milligrams (mg) loading dose in Cycle 1, followed by 420 mg from Cycles 2-4, and docetaxel, 75 milligrams per square meter (mg/m^2) from Cycles 1-4 (1 cycle = 21 days) by intravenous (IV) infusion. Post surgery: Participants received chemotherapy with fluorouracil 500-600 mg/m^2, epirubicin 90-120 mg/m^2, and cyclophosphamide 500-600 mg/m^2 by IV infusion every 3 weeks from Cycles 5-7 (1 cycle = 21 days) followed by trastuzumab, 8 mg/kg loading dose in Cycle 8, followed by 6 mg/kg from Cycles 9-20 and pertuzumab, 840 mg loading dose in Cycle 8, followed by 420 mg from Cycles 9-20 (1 cycle = 21 days).
- Placebo, Trastuzumab, and Chemotherapy: Prior to surgery: Participants received trastuzumab, 8 mg/kg loading dose in Cycle 1, followed by 6 mg/kg from Cycles 2-4, docetaxel, 75 mg/m^2 and placebo from Cycles 1-4 (1 cycle = 21 days) by IV infusion. Post surgery: Participants received chemotherapy with fluorouracil 500-600 mg/m^2, epirubicin 90-120 mg/m^2, and cyclophosphamide 500-600 mg/m^2 by IV infusion every 3 weeks from Cycles 5-7 (1 cycle = 21 days) followed by trastuzumab, 8 mg/kg loading dose in Cycle 8, followed by 6 mg/kg from Cycles 9-20 and placebo from Cycles 8-20 (1 cycle =21 days).
Period: Neoadjuvant Treatment
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Started (Intent-to-Treat (ITT) Population) | 219 | 110
Received at Least One Dose of Study Treatment (Safety Evaluable Population) | 218 | 110
Completed Neoadjuvant Treatment | 214 | 108
Underwent Surgery | 210 | 105
Completed | 208 | 103
Not Completed | 11 | 7
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Progression of Disease | 2 | 3
Not completed — Did Not Receive Study Drug | 1 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 2 | 1
Period: Adjuvant Treatment
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Started | 208 | 103
Started Adjuvant FEC Treatment | 208 | 103
Started Adjuvant Anti-HER2 Treatment | 204 | 99
Completed (Completed Adjuvant anti-HER2 Treatment) | 198 | 94
Not Completed | 10 | 9
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Recurrent Disease | 4 | 5
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 1 | 0
Period: Treatment-Free Follow-Up
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Started (Includes those who had discontinued from neoadjuvant and/or adjuvant treatment but remained in follow-up.) | 208 | 104
Completed | 175 | 82
Not Completed | 33 | 22
Not completed — Death | 11 | 11
Not completed — Lost to Follow-up | 9 | 4
Not completed — Withdrawal by Subject | 13 | 3
Not completed — Non-compliance | 0 | 1
Not completed — Reason Not Specified | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) population included all participants who were enrolled regardless of whether they received any study treatment.
Groups:
- Pertuzumab, Trastuzumab, and Chemotherapy: Prior to surgery: Participants received trastuzumab, 8 mg/kg loading dose in Cycle 1, followed by 6 mg/kg from Cycles 2-4, pertuzumab, 840 mg loading dose in Cycle 1, followed by 420 mg from Cycles 2-4, and docetaxel, 75 mg/m^2 from Cycles 1-4 (1 cycle = 21 days) by IV infusion. Post surgery: Participants received chemotherapy with fluorouracil 500-600 mg/m^2, epirubicin 90-120 mg/m^2, and cyclophosphamide 500-600 mg/m^2 by IV infusion every 3 weeks from Cycles 5-7 (1 cycle = 21 days) followed by trastuzumab, 8 mg/kg loading dose in Cycle 8, followed by 6 mg/kg from Cycles 9-20 and pertuzumab, 840 mg loading dose in Cycle 8, followed by 420 mg from Cycles 9-20 (1 cycle = 21 days).
- Total: Total of all reporting groups
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy | Total
Number analyzed (Participants) | 219 | 110 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.7) | 49.5 (9.1) | 48.8 (9.5)
Age, Customized [Count of Participants; unit: Participants]
  <40 years old | 40 | 18 | 58
  40-49 years old | 75 | 40 | 115
  50-64 years old | 96 | 44 | 140
  ≥65 years old | 8 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219 | 110 | 329
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 219 | 110 | 329
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 219 | 110 | 329
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Disease Category [Count of Participants; unit: Participants] — Population: ITT Population
  Participants
    Early Stage | 152 | 77 | 229
    Locally Advanced | 67 | 33 | 100
Hormone Receptor Status [Count of Participants; unit: Participants]
  Estrogen Receptor (ER) and Progesterone Receptor (PgR) Negative | 105 | 54 | 159
  Estrogen Receptor (ER) and/or Progesterone Receptor (PgR) Positive | 114 | 56 | 170
Baseline LVEF value [Mean (Standard Deviation); unit: percentage points of LVEF] — Left ventricular ejection fraction (LVEF) is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. A normal LVEF ranges from 55% to 70%, as measured by echocardiogram or multiple-gated acquisition (MUGA) scan. Population: Safety Evaluable Population; only participants who received at least one dose of study drug are included.
  percentage points of LVEF
    number analyzed (Participants) | 218 | 110 | 328
    (all) | 66.41 (4.93) | 66.03 (5.19) | 66.28 (5.01)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Total Pathologic Complete Response (tpCR) as Assessed by the Independent Review Committee (IRC)
Description: This tpCR was assessed by the IRC. tpCR was defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes after completion of neoadjuvant therapy and surgery (that is, ypT0/is, ypN0, in accordance with the current American Joint Committee on Cancer [AJCC] staging system). The analysis was based on the ITT population with participants grouped by the treatment assigned at the time of randomization. Participants whose tpCR assessment was missing or invalid were counted as not achieving tpCR. The duration of one treatment cycle was 21 days; the administration of therapy in Cycle 5 did not occur until 2 weeks after surgery. The percentages have been rounded off to first decimal point.
Time Frame: At surgery (Cycle 4 Days 22-35)
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
percentage of participants | 39.3 [32.76 to 46.08] | 21.8 [14.51 to 30.70]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Test type: Superiority; p = 0.0014, Cochran-Mantel-Haenszel — Two-sided significance level of 5%; Stratified by disease category (early-stage and locally advanced) and hormone-receptor status (positive for ER and/or PgR or negative for both); Difference in response rates = 17.45, 95% CI 2-sided [6.89 to 28.01] — Pertuzumab, Trastuzumab, Docetaxel arm minus Placebo, Trastuzumab, Docetaxel arm. Approximate 95% CI for difference of two rates using Hauck-Anderson method

2. Secondary Outcome: Percentage of Participants With tpCR as Assessed by the Local Pathologist
Description: This tpCR was assessed by the local pathologist. tpCR was defined as the absence of any residual invasive cancer on hematoxylin and eosin evaluation of the resected breast specimen and all sampled ipsilateral lymph nodes after completion of neoadjuvant therapy and surgery (that is, ypT0/is, ypN0, in accordance with the current AJCC staging system). The analysis was based on the ITT population with participants grouped by the treatment assigned at the time of randomization. Participants whose tpCR assessment was missing or invalid were counted as not achieving tpCR. The duration of one treatment cycle was 21 days; the administration of therapy in Cycle 5 did not occur until 2 weeks after surgery. The percentages have been rounded off to first decimal point.
Time Frame: At surgery (Cycle 4 Days 22-35)
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
percentage of participants | 39.3 [32.76 to 46.08] | 20.9 [13.74 to 29.70]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — Two-sided significance level of 5%; [statistical method as in outcome 1, analysis 1]; Difference in response rates = 18.36, 95% CI 2-sided [7.89 to 28.83] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With Breast Pathologic Complete Response (bpCR), Defined as ypT0/is According to the AJCC Staging System as Assessed by the IRC
Description: This bpCR was assessed by the IRC. bpCR was defined as the absence of any residual invasive cancer on the hematoxylin and eosin evaluation of the resected breast specimen after completion of neoadjuvant therapy and surgery (that is, ypT0/is, in accordance with current AJCC staging system). The analysis was based on the ITT population with participants grouped by the treatment assigned at the time of randomization. Participants whose bpCR assessment was missing or invalid were counted as not achieving bpCR. The duration of one treatment cycle was 21 days; the administration of therapy in Cycle 5 did not occur until 2 weeks after surgery. The percentages have been rounded off to first decimal point.
Time Frame: At surgery (Cycle 4 Days 22-35)
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Pertuzumab, Trastuzumab, and Chemotherapy: Prior to surgery: Participants received trastuzumab, 8 mg/kg loading dose in Cycle 1, followed by 6 mg/kg from Cycles 2-4, pertuzumab, 840 mg loading dose in Cycle 1, followed by 420 mg from Cycles 2-4, and docetaxel 75 mg/m^2 from Cycles 1-4 (1 cycle = 21 days) by IV infusion. Post surgery: Participants received chemotherapy with fluorouracil 500-600 mg/m^2, epirubicin 90-120 mg/m^2, and cyclophosphamide 500-600 mg/m^2 by IV infusion every 3 weeks from Cycles 5-7 (1 cycle = 21 days) followed by trastuzumab, 8 mg/kg loading dose in Cycle 8, followed by 6 mg/kg from Cycles 9-20 and pertuzumab, 840 mg loading dose in Cycle 8, followed by 420 mg from Cycles 9-20 (1 cycle = 21 days).
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
percentage of participants | 42.0 [35.39 to 48.85] | 23.6 [16.06 to 32.68]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel — Two-sided significance level of 5%; [statistical method as in outcome 1, analysis 1]; Difference in response rates = 18.37, 95% CI 2-sided [7.60 to 29.15] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Percentage of Participants With bpCR as Assessed by the Local Pathologist
Description: This bpCR was assessed by the local pathologist. bpCR was defined as the absence of any residual invasive cancer on the hematoxylin and eosin evaluation of the resected breast specimen after completion of neoadjuvant therapy and surgery (that is, ypT0/is in accordance with current AJCC staging system). The analysis was based on the ITT population with participants grouped by the treatment assigned at the time of randomization. Participants whose bpCR assessment was missing or invalid were counted as not achieving bpCR. The duration of one treatment cycle was 21 days; the administration of therapy in Cycle 5 did not occur until 2 weeks after surgery. The percentages have been rounded off to first decimal point.
Time Frame: At surgery (Cycle 4 Days 22-35)
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
percentage of participants | 41.6 [34.95 to 48.39] | 22.7 [15.28 to 31.70]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel — Two-sided significance level of 5%; [statistical method as in outcome 1, analysis 1]; Difference in response rates = 18.83, 95% CI 2-sided [8.14 to 29.51] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD) During Cycles 1-4, According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: Clinical responses that include percentage of participants with a CR, PR, SD, or PD were determined by investigator during Cycles 1-4 (prior to surgery) on basis of RECIST version 1.1. CR=disappearance of all target lesions i.e., any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. SD=neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum during the study. PD=at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (nadir) with inclusion of baseline. Only participants with measurable disease at baseline were included in the analysis. 1 Cycle=21 days. The percentages have been rounded off to first decimal point.
Time Frame: At surgery (Cycle 4 Days 22-35)
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
percentage of participants
  Complete Response | 11.0 [7.15 to 15.87] | 10.0 [5.10 to 17.19]
  Partial Response | 77.6 [71.52 to 82.97] | 68.2 [58.62 to 76.74]
  Stable Disease | 8.2 [4.94 to 12.68] | 19.1 [12.22 to 27.69]
  Progressive Disease | 0.5 [0.01 to 2.52] | 1.8 [0.22 to 6.41]
  Missing or Unevaluable | 2.7 [NA to NA] — 95% confidence intervals were only calculated for clinical responses. | 0.9 [NA to NA] — 95% confidence intervals were only calculated for clinical responses.

6. Secondary Outcome: Percentage of Participants With an Objective Response (CR or PR) During Cycles 1-4, According to RECIST Version 1.1
Description: An objective response was defined as the percentage of participants who achieved a CR or PR as the best tumor response during the neoadjuvant period (that is, during Cycles 1-4 prior to surgery), as determined by the investigator on the basis of RECIST version 1.1. CR=disappearance of all target lesions i.e., any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR=at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters. No confirmation was required for objective response. Only participants with measurable disease at baseline were included in the analysis. The duration of one treatment cycle was 21 days; the administration of therapy in Cycle 5 did not occur until 2 weeks after surgery. The percentages have been rounded off to first decimal point.
Time Frame: At surgery (Cycle 4 Days 22-35)
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
percentage of participants | 88.6 [83.61 to 92.47] | 78.2 [69.30 to 85.49]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Test type: Superiority; p = 0.0125, Cochran-Mantel-Haenszel — Two-sided significance level of 5%; [statistical method as in outcome 1, analysis 1]; Difference in response rates = 10.40, 95% CI 2-sided [1.12 to 19.69] — Pertuzumab, Trastuzumab, Docetaxel arm minus Placebo, Trastuzumab, Docetaxel arm

7. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Event-Free Survival (EFS) at 1, 3, and 5 Years
Description: Kaplan-Meier approach was used to estimate percentage of participants who were event-free for EFS at 1, 3 & 5 years. EFS=time from randomization to first documentation of one of the following events: PD (before surgery) as determined by investigator with RECIST v1.1. PD=at least a 20% increase in sum of diameters of target lesions, taking as reference smallest sum during the study (nadir) with inclusion of baseline. Any evidence of contralateral disease in situ was not identified as PD; Disease recurrence (local, regional, distant, or contralateral) after surgery; Death from any cause. After treatment completion/discontinuation, follow-up data was collected every 3 months for 1 year & then every 6 months thereafter, until disease progression/recurrence or until 5 years after randomization of last participant, whichever occurred first. Participants without an EFS event at time of analysis were censored as of the date they were last known to be alive & event-free.
Time Frame: From Baseline to EFS event or date last known to be alive and event-free at 1, 3, and 5 years
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an EFS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: estimate of percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
estimate of percentage of participants
  1 Year: number analyzed (Participants) | 204 | 93
  1 Year | 98.62 [97.06 to 100.00] | 90.46 [84.82 to 96.09]
  3 Years: number analyzed (Participants) | 176 | 80
  3 Years | 88.85 [84.55 to 93.15] | 79.68 [71.91 to 87.45]
  5 Years: number analyzed (Participants) | 151 | 67
  5 Years | 84.80 [79.86 to 89.73] | 73.70 [65.17 to 82.23]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Hazard Ratio for EFS Event in the Pertuzumab arm vs. Placebo arm; Test type: Superiority; p = 0.0140, Stratified log-rank; Two-sided log-rank test used, stratified by disease category (early-stage/locally advanced) & hormone-receptor status (ER+ &/or PgR+ or ER- & PgR-); Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.32 to 0.89] — The hazard ratio was calculated by stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in EFS Event-Free Rates at 1 year; Test type: Superiority; p = 0.0062, Z-test; Difference in EFS Event-Free Rates = -8.16, 95% CI 2-sided [-14.00 to -2.32] — The difference in EFS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm
Statistical Analysis 3: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in EFS Event-Free Rates at 3 years; Test type: Superiority; p = 0.0429, Z-test; Difference in EFS Event-Free Rates = -9.17, 95% CI 2-sided [-18.05 to -0.29] — The difference in EFS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm
Statistical Analysis 4: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in EFS Event-Free Rates at 5 Years; Test type: Superiority; p = 0.0274, Z-test; Difference in EFS Event-Free Rates = -11.10, 95% CI 2-sided [-20.95 to -1.24] — The difference in EFS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm

8. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Disease-Free Survival (DFS) at 1, 3, and 5 Years
Description: Kaplan-Meier approach was used to estimate the percentage of participants who were event-free for DFS at 1, 3 and 5 years. DFS = time from first date of no disease (i.e., date of surgery) to first documentation of one of the following events: Disease recurrence (local, regional, distant, or contralateral) after surgery or death from any cause. After treatment completion/discontinuation, follow-up data was collected every 3 months for 1 year and then every 6 months thereafter, until disease progression or recurrence or until 5 years after randomization of the last participant, whichever occurred first. Participants were considered to be disease-free if they underwent surgery and no recurrence of disease was reported thereafter. Data from participants who did not have an event at analysis were censored as of the date they were last known to be alive and event-free.
Time Frame: From surgery (Cycle 4: Days 22-35) to DFS event or date last known to be alive and event-free at 1, 3, and 5 years
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment. Overall number of participants analyzed are unique number of participants who underwent surgery. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for a DFS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: estimate of percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 210 | 105
estimate of percentage of participants
  1 Year: number analyzed (Participants) | 197 | 93
  1 Year | 97.55 [95.42 to 99.67] | 92.08 [86.81 to 97.35]
  3 Years: number analyzed (Participants) | 176 | 80
  3 Years | 90.09 [85.97 to 94.22] | 81.10 [73.44 to 88.75]
  5 Years: number analyzed (Participants) | 81 | 41
  5 Years | 85.99 [81.17 to 90.80] | 75.02 [66.53 to 83.51]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Hazard Ratio for DFS Event in the Pertuzumab arm vs. Placebo arm; Test type: Superiority; p = 0.0140, Stratified log-rank; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.30 to 0.88] — The hazard ratio was calculated by stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in DFS Event-Free Rates at 1 year; Test type: Superiority; p = 0.0592, Z-test; Difference in DFS Event-Free Rates = -5.47, 95% CI 2-sided [-11.15 to 0.21] — The difference in DFS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm
Statistical Analysis 3: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in DFS Event-Free Rates at 3 years; Test type: Superiority; p = 0.0426, Z-test; Difference in DFS Event-Free Rates = -9.00, 95% CI 2-sided [-17.69 to -0.30] — The difference in DFS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm
Statistical Analysis 4: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in DFS Event-Free Rates at 5 years; Test type: Superiority; p = 0.0276, Z-test; Difference in DFS Event-Free Rates = -10.97, 95% CI 2-sided [-20.73 to -1.21] — The difference in DFS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm

9. Secondary Outcome: Kaplan-Meier Estimate of the Percentage of Participants Event-Free for Overall Survival (OS) at 1, 3, and 5 Years
Description: Kaplan-Meier approach was used to estimate the percentage of participants who were event-free for OS at 1, 3 and 5 years. OS was defined as the time from randomization to death from any cause. After treatment completion/discontinuation, follow-up data was collected every 3 months for 1 year and then every 6 months thereafter, until disease progression or recurrence or until 5 years after randomization of the last participant, whichever occurred first. Data from participants who were alive at the time of the analysis was censored as of the last date they were known to be alive.
Time Frame: From Baseline to OS event or date last known to be alive at 1, 3, and 5 years
Population: ITT population included all participants who were enrolled regardless of whether they received any study treatment. Number analyzed per timepoint are unique number of participants out of all the assessed participants who remain at risk for an OS event at that timepoint. Different participants may have contributed data for each timepoint.
Measure: Number (95% Confidence Interval); unit: estimate of percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 219 | 110
estimate of percentage of participants
  1 Year: number analyzed (Participants) | 205 | 101
  1 Year | 99.54 [98.64 to 100.00] | 100.00 [100.00 to 100.00]
  3 Years: number analyzed (Participants) | 188 | 89
  3 Years | 97.01 [94.64 to 99.37] | 90.99 [85.37 to 96.60]
  5 Years: number analyzed (Participants) | 160 | 77
  5 Years | 93.86 [90.49 to 97.23] | 89.97 [84.06 to 95.87]
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Hazard Ratio for OS Event in the Pertuzumab arm vs. Placebo arm; Test type: Superiority; p = 0.1181, Stratified log-rank; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.23 to 1.19] — The hazard ratio was calculated by stratified Cox proportional hazards model
Statistical Analysis 2: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in OS Event-Free Rates at 1 year; Test type: Superiority; p = 0.3162, Z-test; Difference in OS Event-Free Rates = 0.46, 95% CI 2-sided [-0.44 to 1.36] — The difference in OS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm
Statistical Analysis 3: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in OS Event-Free Rates at 3 years; Test type: Superiority; p = 0.0529, Z-test; Difference in OS Event-Free Rates = -6.02, 95% CI 2-sided [-12.11 to 0.08] — The difference in OS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm
Statistical Analysis 4: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Difference in OS Event-Free Rates at 5 years; Test type: Superiority; p = 0.2616, Z-test; Difference in OS Event-Free Rates = -3.89, 95% CI 2-sided [-10.69 to 2.90] — The difference in OS event-free rates was calculated as the Placebo arm minus the Pertuzumab arm

10. Secondary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During the Neoadjuvant Treatment Period
Description: The percentage of participants who experienced at least one AE during the neoadjuvant period is reported here. An AE is any untoward medical occurrence in a clinical investigation participant who is administered a pharmaceutical product regardless of the causal attribution. An adverse event was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsened during the study were also considered as adverse events. The neoadjuvant treatment period began after randomization upon receiving the first dose of any of the neoadjuvant study medications and ended before receiving the first dose of adjuvant study treatment. The duration of one treatment cycle is 21 days. The percentages have been rounded off to first decimal point.
Time Frame: Baseline up to end of Cycle 4 (1 cycle = 21 days)
Population: Safety evaluable population included all participants who received at least one dose of neoadjuvant study treatment and participants were grouped by the treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 218 | 110
percentage of participants | 97.7 | 96.4

11. Secondary Outcome: Percentage of Participants With at Least One AE During the Adjuvant Treatment Period
Description: Percentage of participants who experienced at least one adverse event during the adjuvant period is reported here. An AE is any untoward medical occurrence in a clinical investigation participant who is administered a pharmaceutical product regardless of the causal attribution. An adverse event was therefore any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Pre-existing conditions which worsened during the study were also considered as adverse events. Adjuvant treatment period began after primary surgery, upon receiving the first dose of any of the adjuvant study medications. It ended 42 days after last dose of adjuvant study treatment upon treatment completion or discontinuation. 1 Cycle=21 days. The percentages have been rounded off to first decimal point.
Time Frame: From Cycle 5 (1 cycle = 21 days) up to 42 days after the last dose in Cycle 20 Day 1 (approximately 1 year)
Population: Safety evaluable population included all participants who received at least one dose of adjuvant study treatment and participants were grouped by the treatment they actually received. Overall number analyzed is the number of participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 208 | 103
percentage of participants | 98.1 | 98.1

12. Secondary Outcome: Percentage of Participants With at Least One Adverse Event During the Treatment-Free Follow-Up Period
Description: The percentage of participants who experienced at least one adverse event during the treatment-free follow-up period is reported here. An AE is any untoward medical occurrence in a clinical investigation participant who is administered a pharmaceutical product regardless of the causal attribution. An adverse event was therefore any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. The percentages have been rounded off to first decimal point.
Time Frame: From end of overall study treatment until disease progression or until 5 years after randomization of the last patient, whichever occurred first (up to 6 years)
Population: Safety evaluable population included all participants who received at least one dose of study drugs and participants were grouped by the treatment they actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 218 | 110
percentage of participants | 6.0 | 7.3

13. Secondary Outcome: Percentage of Participants Who Experienced a Primary Cardiac Event
Description: A primary cardiac event is defined as heart failure (New York Heart Association [NYHA] Class III or NYHA Class IV) and a drop in left ventricular ejection fraction (LVEF) of at least 10 ejection fraction points from baseline and to below 50%.
Time Frame: From Baseline until end of study (up to 6 years)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 218 | 110
percentage of participants | 0 | 0

14. Secondary Outcome: Percentage of Participants Who Experienced a Secondary Cardiac Event
Description: A secondary cardiac event is defined as an asymptomatic or mildly symptomatic (NYHA Class II) drop in LVEF by multiple-gated acquisition (MUGA) scan or echocardiogram confirmed by a second LVEF assessment within approximately 3 weeks showing also a documented drop. A significant LVEF drop is defined as an absolute decrease of at least 10 points below the baseline measurement and to below 50%.
Time Frame: From Baseline until end of study (up to 6 years)
Population: as for outcome 12
Measure: Number; unit: percentage of participants
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 218 | 110
percentage of participants | 0 | 0

15. Secondary Outcome: Maximum Change From Baseline in LVEF
Description: LVEF is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. A normal LVEF ranges from 55% to 70%, as measured by echocardiogram (preferred) or MUGA scan. The same method was used throughout the study for each participant and preferably performed and evaluated by the same assessor. Here, we report the maximum change from baseline in LVEF at any point during the study.
Time Frame: Baseline; Day 1 of Cycles 2, 4, 5, 8, 11, and 20 (1 cycle = 21 days)
Population: Safety evaluable population included all participants who received at least one dose of study drugs and participants were grouped by the treatment they actually received. Overall number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: percentage points of LVEF
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 215 | 109
percentage points of LVEF | -6.55 (5.22) | -6.20 (6.08)
Statistical Analysis 1: Comparison: Pertuzumab, Trastuzumab, and Chemotherapy vs Placebo, Trastuzumab, and Chemotherapy; Test type: Other; Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-1.62 to 0.93] — Pertuzumab, Trastuzumab, Docetaxel arm minus Placebo, Trastuzumab, Docetaxel arm

16. Secondary Outcome: Change From Baseline in LVEF Over Time
Description: LVEF is the measurement of how much blood is being pumped out of the left ventricle of the heart (the main pumping chamber) with each contraction. A normal LVEF ranges from 55% to 70%, as measured by echocardiogram (preferred) or MUGA scan. The same method was used throughout the study for each participant and preferably performed and evaluated by the same assessor. Here, we report the change from baseline in LVEF over time.
Time Frame: Baseline; Day 1 of Cycles 2, 4, 5, 8, 11, and 20 (1 cycle = 21 days)
Population: Safety evaluable population included all participants who received at least one dose of study drugs. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at specified timepoints.
Measure: Mean (95% Confidence Interval); unit: percentage points of LVEF
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
Number analyzed (Participants) | 213 | 108
percentage points of LVEF
  Cycle 2 Day 1 | -0.62 [-1.35 to 0.11] | 0.29 [-0.89 to 1.46]
  Cycle 4 Day 1: number analyzed (Participants) | 212 | 108
  Cycle 4 Day 1 | -1.02 [-1.72 to -0.32] | 0.09 [-1.03 to 1.22]
  Cycle 5 Day 1: number analyzed (Participants) | 200 | 102
  Cycle 5 Day 1 | -0.96 [-1.70 to -0.22] | 0.07 [-1.12 to 1.26]
  Cycle 8 Day 1: number analyzed (Participants) | 196 | 97
  Cycle 8 Day 1 | -1.63 [-2.44 to -0.81] | -1.18 [-2.30 to -0.05]
  Cycle 11 Day 1: number analyzed (Participants) | 203 | 94
  Cycle 11 Day 1 | -1.38 [-2.16 to -0.61] | -0.65 [-1.91 to 0.62]
  Cycle 20 Day 1: number analyzed (Participants) | 183 | 89
  Cycle 20 Day 1 | -1.22 [-2.05 to -0.38] | -1.18 [-2.56 to 0.20]

ADVERSE EVENTS:
Time Frame: From first dose of any study drug through end of study (up to 6 years)
Description: Safety Evaluable Population included all participants who received at least one dose of study drugs and participants were grouped by the treatment they actually received. One participant in the pertuzumab arm discontinued from the study before receiving study treatment due to not meeting eligibility criteria. Therefore, there are only 218 participants in the pertuzumab arm in the safety population.
Arm/Group | Pertuzumab, Trastuzumab, and Chemotherapy | Placebo, Trastuzumab, and Chemotherapy
All-Cause Mortality (participants affected / at risk) | 12/218 | 11/110
Serious Adverse Events (participants affected / at risk) | 37/218 | 15/110
Other Adverse Events (participants affected / at risk) | 218/218 | 108/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab, Trastuzumab, and Chemotherapy (N=218) | Placebo, Trastuzumab, and Chemotherapy (N=110)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Blood Loss Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 9 (9) | 3 (3)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelosuppression (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (2) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver Disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver Injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1)
Lung Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 1 (3)
Pneumonia Influenzal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Flap Necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Adnexa Uteri Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Lung Cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abortion Induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Lymphorrhoea (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pertuzumab, Trastuzumab, and Chemotherapy (N=218) | Placebo, Trastuzumab, and Chemotherapy (N=110)
Anaemia (Blood and lymphatic system disorders) | 75 (124) | 36 (66)
Leukopenia (Blood and lymphatic system disorders) | 135 (379) | 67 (160)
Neutropenia (Blood and lymphatic system disorders) | 153 (365) | 73 (161)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (50) | 17 (29)
Abdominal Discomfort (Gastrointestinal disorders) | 11 (11) | 3 (3)
Abdominal Pain Upper (Gastrointestinal disorders) | 11 (11) | 8 (8)
Constipation (Gastrointestinal disorders) | 25 (26) | 15 (21)
Diarrhoea (Gastrointestinal disorders) | 87 (124) | 19 (20)
Mouth Ulceration (Gastrointestinal disorders) | 30 (38) | 10 (10)
Nausea (Gastrointestinal disorders) | 84 (147) | 40 (69)
Stomatitis (Gastrointestinal disorders) | 7 (10) | 7 (8)
Vomiting (Gastrointestinal disorders) | 36 (47) | 13 (17)
Asthenia (General disorders) | 19 (22) | 8 (9)
Chills (General disorders) | 12 (13) | 3 (4)
Fatigue (General disorders) | 26 (42) | 16 (26)
Malaise (General disorders) | 13 (14) | 5 (7)
Oedema Peripheral (General disorders) | 11 (14) | 8 (8)
Pyrexia (General disorders) | 37 (47) | 16 (17)
Hepatic Function Abnormal (Hepatobiliary disorders) | 18 (22) | 7 (9)
Nasopharyngitis (Infections and infestations) | 18 (26) | 5 (6)
Upper Respiratory Tract Infection (Infections and infestations) | 58 (85) | 14 (23)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 11 (12) | 3 (3)
Procedural Pain (Injury, poisoning and procedural complications) | 12 (14) | 5 (6)
Radiation Skin Injury (Injury, poisoning and procedural complications) | 23 (23) | 6 (6)
Alanine Aminotransferase Increased (Investigations) | 64 (126) | 41 (62)
Aspartate Aminotransferase Increased (Investigations) | 54 (104) | 34 (48)
Blood Cholesterol Increased (Investigations) | 3 (4) | 6 (6)
Blood Triglycerides Increased (Investigations) | 3 (5) | 7 (17)
Blood Uric Acid Increased (Investigations) | 3 (5) | 8 (13)
Gamma-Glutamyltransferase Increased (Investigations) | 9 (10) | 9 (14)
Low Density Lipoprotein Increased (Investigations) | 5 (5) | 9 (15)
Decreased Appetite (Metabolism and nutrition disorders) | 40 (49) | 13 (19)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (19) | 8 (8)
Bone Pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 9 (10)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 13 (15) | 4 (4)
Dizziness (Nervous system disorders) | 19 (25) | 9 (10)
Headache (Nervous system disorders) | 15 (18) | 6 (6)
Hypoaesthesia (Nervous system disorders) | 14 (15) | 7 (11)
Neuropathy Peripheral (Nervous system disorders) | 12 (12) | 6 (6)
Insomnia (Psychiatric disorders) | 24 (29) | 17 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 23 (26) | 9 (12)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (16) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 20 (24) | 9 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 115 (162) | 56 (77)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (18) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 28 (29) | 22 (26)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 12 (16) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 4 (4) | 7 (7)
Hypertension (Vascular disorders) | 7 (7) | 9 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT02586025/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT02586025/SAP_001.pdf